CLINICAL TRIAL: NCT06762873
Title: Assessment of Obstructive Sleep Apnea in the Latin American Population and Response to Neuromodulation Therapy to Treat Obstructive Sleep Apnea
Brief Title: Assessment of OSA in Latin American and Response to Neuromod Therapy
Acronym: Trans-Q DISE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lunair Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10081
Record Dates: First submitted 2024-12-06; First posted 2025-01-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trans-Q DISE treated subjects (Experimental)
  Interventions: Diagnostic Test: Drug Induced Sleep Endoscopy with PNS

INTERVENTIONS:
Diagnostic Test: Drug Induced Sleep Endoscopy with PNS — Enrolled subjects will complete an overnight PSG and then undergo a DISE procedure with a 30-minute research period.

SUMMARY:
The purpose of this study is to characterize the upper airway of Latin American subjects who have been diagnosed with moderate/severe obstructive sleep apnea (OSA) and assess response to a neuromodulation therapy to treat OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 years old
2. Subject is willing and able to provide informed consent
3. Subject is geographically stable
4. Subject does not have access to alternative Sleep Disordered Breathing treatments (e.g. oral appliances, and/or behavioral treatments)
5. Subject has an Apnea-Hypopnea Index (AHI) score ≥15 < 100 events per hour on Screening PSGs (under AASM 4%) based on in-lab polysomnography studies

Exclusion Criteria:

1. Subject is currently implanted with another active implantable device.
2. Subject is actively enrolled in another premarket investigational study (medical device or drug) unless approved by Sponsor in writing.
3. Subject is considered vulnerable such as incarcerated or cognitively impaired.
4. Subject is taking opioids, narcotics, sleep or psychotic medications or supplements that in the opinion of the investigator may alter consciousness, the pattern of respiration, sleep architecture, or with known effect on sleep-wake function or alertness.
5. Any reason for which, in the judgment of the investigator, the subject is considered to be a poor study candidate, which may include, but is not limited to: any uncontrolled neurological, medical, social, or psychological problems that could complicate the required procedures and evaluations of the study ((e.g. uncontrolled hypertension, unstable angina, uncompensated heart failure or COPD, major depression, Parkinson's disease, epilepsy)
6. Subject has previous upper respiratory tract (URT) surgery (e.g., uvula, soft palate or tonsils) within 60 days prior to Screening PSG.
7. Subject has a need for chronic supplemental oxygen therapy for any reason or a PaO2 <70 mm Hg
8. Subject has other sleep disorders or sleep hygiene behaviors that confound functional assessments of sleepiness and/or overnight PSG Study outcomes (e.g. Narcolepsy with cataplexy, idiopathic hypersomnolence, insomnia, REM sleep behavior disorder, or sleep movement disorders, such as restless leg syndrome or periodic limb movement, producing sleep disturbances unrelated to OSA.)
9. Subject has severe chronic kidney disease (GFR < 30)
10. Subject has currently excessive use of alcohol, tobacco, caffeine, or recreational drugs.
11. Subject is unwilling or unable to refrain from consumption of alcoholic beverages for 24 hours prior to the start of each PSG study.
12. Subject has a BMI > 40 kg/m2
13. Subject has an active systemic infection
14. If female, subject is pregnant at the time of enrollment or planning to become pregnant during the study time period (must have a negative serum or urine pregnancy test within 14 days prior to enrollment)
15. Subject has a tonsil size 3 or 4 based on the tonsil grading system
16. Subject has documented history of Phrenic nerve palsy or asymmetry of the diaphragm
17. Subject has any trauma to the upper airway that interferes with limited tongue movement or inability to move the tongue, tongue dysfunction, atrophy, hypertrophy, fasciculation, or problems swallowing or speaking
18. Subject has severe mandibular deficiency/retrognathia or syndromic craniofacial abnormalities.
19. Subject has previous surgical resection or radiation therapy for cancer or congenital malformations in the larynx, tongue, or throat.
20. Subject has an oxygen saturation (SaO2) >10% falls index > 15 events per hour on Screening PSGs
21. Subject has >25% central apnea events as a proportion of the sum of apnea and hypopnea events per hour on Screening PSGs (up to 3 patients with CAI+MAI ≥ 25% may be included)
22. Subject has sleep Efficiency < 80%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Understand the difference in response compared to prior U.S. based studies to the response in Latin America. | enrollment to study exit, usually within 3 weeks of screening
  Reviewing phrenic nerve stimulation response to literature of US based population
Use VOTE scoring to characterize the type of upper airway collapse as assessed via DISE. | enrollment to study exit, usually within 3 weeks of screening
  Upper Airway will be characterized using VOTE scoring as assessed by a qualified, trained Independent Reviewer.
Use VOTE scoring and airway opening measurements to characterize the effect of Phrenic Nerve Stimulation and if it is a viable and effective treatment of OSA and correlation to phenotype. | enrollment to study exit, usually within 3 weeks of screening
  In combination with VOTE scoring and airway opening measurements, the effects of phrenic nerve stimulation will be compared across treated patient population.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanatorio Americano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No